CLINICAL TRIAL: NCT07102017
Title: The Impact of Socially Supportive Robotic Intervention on Loneliness, Depression, Self-agency and Well-being in Long-term Care Residents: A Three-Arm Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial of Robotic Support for Enhanced Later Life (RoSELL)
Acronym: RoSELL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jianan Zhao, principle investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: L20250617; school (Other: shanghai jiao tong university)
Record Dates: First submitted 2025-07-21; First posted 2025-08-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Loneliness; Well-Being, Psychological; Depression - Major Depressive Disorder
Keywords: Social isolation; socially assistive robots; loneliness; depression; self-agency; well-being
MeSH Terms: conditions — Psychological Well-Being; Social Isolation; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co-designed robot group (Experimental): This intervention arm involves a proactive companion robot delivered over 16 sessions, with a core emphasis on structured personalization to foster attachment.
  Sessions 1-2 (Personalization Ritual): A healthcare professional facilitates a structured, four-phase co-design ceremony.
  Sessions 3-16 (Autonomous Interaction): The co-designed robot is placed in the participant's room for autonomous interaction. It uses the personalized settings and exhibits default affectionate behaviors (e.g., approaching, responding to touch). To reinforce the bond, the healthcare professional uses scripted phrases attributing agency and memory to the robot (e.g., "[Robot's Name] remembers you"). Participants are encouraged to add one new "memory" per session for the robot to "store."
  Interventions: Device: Co-Design LOVOT Intervention
- Standard Robot Group (Experimental): This arm involves the same robot for an equivalent duration and number of sessions as the co-design intervention arm, but without the personalization ritual or anthropomorphic framing.
  Sessions 1-2 (Standardized Introduction): A healthcare professional introduces the same robot, demonstrating its three core, pre-programmed functionalities. The robot has a generic, fixed configuration with identical, pre-set eye color and voice pitch for all participants in this arm.
  Sessions 3-16 (Neutral, Autonomous Interaction): The standard robot is placed in the participant's room for autonomous interaction. The key differentiator is the deliberately neutral and non-anthropomorphic framing by the healthcare professional
  Interventions: Device: Standard LOVOT Intervention
- Control (No Intervention): All groups will receive the usual community center services. The study district offers standard community-based programming, including group exercises, social events, and recreational activities, all of which are accessible to all residents. Participation is voluntary. To control for attention bias, healthcare professionals will conduct weekly 20-minute individual visits with participants in this group, totaling 16 sessions over the 4-week intervention period.

INTERVENTIONS:
Device: Co-Design LOVOT Intervention — This arm utilizes the LOVOT robot within a structured protocol designed to foster a unique personal attachment through a co-design ceremony and anthropomorphic framing.
  Personalization Ritual (Sessions 1-2): A healthcare professional facilitates a multi-phase personalization ceremony.
  Autonomous Interaction (Sessions 3-16): The personalized LOVOT is placed in the participant's room. The robot consistently uses the participant-chosen voice and eye settings.
  Arms: Co-designed robot group
Device: Standard LOVOT Intervention — This arm uses the identical LOVOT robot for an equivalent duration but deliberately excludes personalization and anthropomorphic framing to isolate the effect of generic robot companionship.
  Standardized Introduction (Sessions 1-2): A healthcare professional introduces the LOVOT robot with a fixed, generic configuration.
  Neutral Autonomous Interaction (Sessions 3-16): The standard LOVOT is placed in the participant's room. The robot operates with its default outgoing personality and identical sensors (thermal camera, touch, distance) for safe, autonomous movement and recharging.
  Arms: Standard Robot Group

SUMMARY:
The purpose of this study is to compare the efficacy of a personalized, co-designed robot interaction against a standardized, fixed robot interaction for reducing loneliness, depression, as well as improving self-agency and quality of life in older adults.

This is a three-arm randomized controlled trial. The study will be conducted at a community center in Fuzhou, China, with 100 participants aged 65+ recruited from the facility. The participants will be randomly assigned to one of three conditions: (1) Co-designed robot (CL) group receiving a personalized robot interaction with a structured co-design ceremony; (2) Standard robot (SL) group interacting with an identical robot without personalization features; or (3) An attention-controlled usual care (CU) group. The intervention comprises 16 sessions (two weekly 20-minute sessions over eight weeks). The primary outcomes are loneliness and depressive symptoms. Secondary outcomes include general self-efficacy, quality of life, as well as staff and participants' perceptions of the robot. Mechanism measures (i.e., engagement, self-disclosure) and manipulation checks (e.g., perceived personal role) will be employed to elucidate the underlying theoretical pathways. Data will be collected at baseline (T0), after the initial 2-week co-design period (T1), post-intervention (T2, Week 8), and at 1-month (T3) and 3-month (T4) follow-ups.

ELIGIBILITY:
The inclusion criteria of this program are: (1) being aged 65 or above, (2) living within the elderly community center for at least 1 month, and (3) being capable of interacting with a robot.

The participants were not eligible if they were: (1) already engaged in other socially assistive robot programs, (2) diagnosed with severe psychiatric problems, (3) bed-bound, or (4) living in an area with no Internet coverage.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Loneliness | From enrollment to the end of treatment at 24 weeks
  Measure the loneliness of participants at baseline before the intervention (T0), at the end of Week 2 (T1) following the initial interaction period, at the end of Week 8 (T2) upon completion of the core intervention phase, and at Week 12 (T3) and Week 24 (T4) to assess the sustained effects of the intervention.
Depression | From enrollment to the end of treatment at 24 weeks.
  Depressive Symptoms will be assessed using the Chinese version of the 15-item Geriatric Depression Scale (GDS-15) at baseline before the intervention (T0), at the end of Week 2 (T1) following the initial interaction period, at the end of Week 8 (T2) upon completion of the core intervention phase, and at Week 12 (T3) and Week 24 (T4).

SECONDARY OUTCOMES:
Self-Efficacy | From enrollment to the end of treatment at 24 weeks
  General Self-Efficacy will be measured by the Chinese version of the General Self-Efficacy Scale (GSES) at baseline before the intervention (T0), at the end of Week 2 (T1) following the initial interaction period, at the end of Week 8 (T2) upon completion of the core intervention phase, and at Week 12 (T3) and Week 24 (T4).
Quality of life and Wellbeing | From enrollment to the end of treatment at 24 weeks
  Quality of Life will be evaluated using the WHO-5 Well-Being Index at baseline before the intervention (T0), at the end of Week 2 (T1) following the initial interaction period, at the end of Week 8 (T2) upon completion of the core intervention phase, and at Week 12 (T3) and Week 24 (T4).

OTHER OUTCOMES:
Interaction engagement | From enrollment to the end of treatment at 8 weeks
  The degree of engagement experienced during interactions will be captured using a scale that measures the level of absorption and focused engagement with the robot at pre- and post-intervention time points (T1, T2)
Self-disclosure | From enrollment to the end of treatment at 8 weeks.
  Participants' intention of sharing personal information, thoughts, feelings, and experiences when interacting with the robot will be evaluated through a measure of self-disclosure specific to the human-robot interaction context at pre-intervention and post-intervention time points (T1, T2).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
For protecting user privacy